CLINICAL TRIAL: NCT03792113
Title: EVALUATION AND COMPARISON OF THE EFFICACY OF AUTOLOGOUS FIBRIN GLUE WITH 4-0 SILK SUTURES IN PERIODONTAL FLAP CLOSURE AND WOUND HEALING - A SPLIT MOUTH RANDOMIZED CONTROLLED TRIAL.
Brief Title: AUTOLOGOUS FIBRIN GLUE VERSES 4-0 SILK SUTURES IN PERIODONTAL FLAP CLOSURE
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: KLE Society's Institute of Dental Sciences (Other)
Responsible Party: Principal Investigator, Dr Laveena Singhal, Post graduate student, Principal investigator, Department of Periodontics, KLE Society's Institute of Dental Sciences, Bangalore, KLE Society's Institute of Dental Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: nehafibringlue
Record Dates: First submitted 2019-01-01; First posted 2019-01-03 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Intervention Model Description: Patients diagnosed with periodontitis, in the age group of 18 to 60 years with good systemic health and presence of a minimum of 3 teeth with periodontal pocket depth (PPD) of ≥6mm and clinical attachment level (CAL) of ≥5mm
Who Masked: Investigator, Outcomes Assessor
Masking Description: The study design follows a double blinded design where the investigator and the outcome assessor are unaware of the intervention to the subject
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Autologous fibrin glue (Experimental): The periodontal flap will be approximated on the test site using autologous fibrin glue on the under surface of the raised flap up to 2 mm from the coronal margin and repositioned back on to the root surface. Thereafter, the tissues will be kept in position with a gentle pressure using a wet gauze for 30 - 60 seconds.
  Interventions: Procedure: Periodontal Flap Surgery; Other: Autologous fibrin glue
- 4-0 silk suture (Active Comparator): The periodontal flap will be approximated using 4-0 black silk suture.
  Interventions: Procedure: Periodontal Flap Surgery; Other: 4-0 silk suture

INTERVENTIONS:
Procedure: Periodontal Flap Surgery — Periodontal access flap surgery will be performed in both test site followed by control site in each subject
Other: Autologous fibrin glue — Autologous fibrin glue procured from the subject's own venous blood will be used to approximate periodontal flaps following access periodontal surgery
  Arms: Autologous fibrin glue
Other: 4-0 silk suture — Conventional 4-0 black silk suture will be used to approximate periodontal flaps following access flap surgery
  Arms: 4-0 silk suture

SUMMARY:
The study is a split mouth study but the interventions for the two different arms will be spaced by a fixed duration in time. Verbal and written consent will be obtained from the patients fulfilling the inclusion and exclusion criteria after briefing them about the procedure. Following phase-1 periodontal therapy, randomisation for the test and control quadrants will be done. Surgical debridement will be done first for the control side to avoid the carry-across effect of fibrin glue. Control and test procedures will be performed with a wash out period of 15days.

Preparation of Autologous fibrin glue :

* 10 ml of blood will be withdrawn from healthy adult human donor by venous puncture into sodium citrate vials and will be centrifuged for 30 min at 1200 g to obtain platelet-poor plasma (PPP).
* To the solution, fibrinogen and protamine sulphate will be added and will be centrifuged at 1000 g for 5 min to sediment the precipitate and fibrin glue will be procured.

Prior to commencement of periodontal flap surgery GCF collection will be done. Following anaesthesia and elevation of full thickness muco periosteal flap, thorough debridement and root planning of the exposed root surfaces will be done. On the control site, the periodontal flap will be approximated using 4-0 black silk suture. Patients will be instructed to rinse twice daily with 0.12% chlorhexidine and recalled after 7 days for suture removal and post-surgical GCF collection from the control side. After a wash out period of 15 days presurgical GCF sampling along with the surgical procedure will be performed on the test side. The periodontal flap will be approximated on the test site using autologous fibrin glue on the under surface of the raised flap up to 2 mm from the coronal margin and repositioned back on to the root surface. Thereafter, the tissues will be kept in position with a gentle pressure using a wet gauze for 30 - 60 seconds. Persistence of bleeding, stability of tissues 5 minutes after repositioning will be recorded and the amount of fibrin sealant used in the procedure will be determined.Patients will be then recalled after 7 days for evaluation and post-surgical GCF collection from the test site. Clinical parameters will be assessed at 7, 14, 21 and 28 days.

Collection of GCF :

GCF will be collected immediately prior to surgery and on seventh day following surgery from both test and control sites for wound healing assessment. Samples of GCF will be collected from four sites from the surgical site following isolation. Colour - coded, 1-5 microlitre calibrated volumetric micro capillary pipettes will be kept extra-crevicularly for not more than five minutes or until 1 microlitre is collected. The fluid will be immediately transferred to a plastic vial and frozen at -20 degree Celsius for further analysis. Pipettes in sites which do not express any fluid or those contaminated with blood/saliva will be discarded.

Statistical analysis:

The data gathered from the study will be subjected to appropriate statistical analysis. The statistical analysis will be done using:

1. Mann-Whitney test
2. Wilcoxon signed rank test.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with periodontitis, with good systemic health and presence of a minimum of 3 teeth with periodontal pocket depth (PPD) of ≥6mm and clinical attachment level (CAL) of ≥5mm (stage 3 periodontitis as described by the 2017 World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Condition and published by the American Academy of Periodontology) in at least two quadrants will be selected.

Exclusion Criteria:

* Patients who have undergone periodontal therapy during the previous 6 months, or exhibit poor plaque control after phase I therapy.
* History of any systemic disease such as diabetes mellitus, hypertension,osteoporosis, unstable or life-threatening conditions, bleeding disorder, undergoing antibiotic or other antimicrobial therapy.
* Patients on drugs like aspirin, blood thinners and anticoagulant therapy
* Patients with history of allergy
* Current or former smokers.
* Mobility of selected teeth.
* Pregnant or lactating women.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-05 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Cytokine parameter | Change from baseline to 7days
  Interleukin 1-β will be assessed in GCF using a commercially available Enzyme-linked immunosorbent assay kit (ELISA), specific for human IL-1 β

SECONDARY OUTCOMES:
Oral Hygiene Index | Changes from baseline to 7day, 14day, 21day, 28day
  by John C Greene & Jack Vermilion in 1964 OHI = DI + CI INTERPRETATION Good 0.0-1.2 Fair 1.3-3.0 Poor 3.1-6.0
Early Wound Healing Index | Changes from baseline to 7th day, 14th day, 21st day and 28th day
  Index given by Watchel et al in 2005
  SCORING CRITERIA:
  DEGREE 1-Complete flap closure No fibrin line in the interproximal area DEGREE 2- Complete flap closure Fine fibrin line in the interproximal area DEGREE 3- Complete flap closure Fibrin clot in the interproximal area DEGREE 4- Incomplete flap closure Partial necrosis of interproximal tissue DEGREE 5- Incomplete flap closure Complete necrosis of interproximal tissue
Gingival Index | Changes from baseline to 7th day, 14th day, 21st day and 28th day
  Index given by Loe and Silness in 1963 Scoring criteria 0 = Normal gingiva
  1. = Mild inflammation, slight change in color, slight edema, no bleeding on probing.
  2. = Moderate inflammation, redness, edema, and glazing, bleeding on probing.
  3. = Severe inflammation, marked redness and edema, ulceration, tendency to spontaneous bleeding.
  Score 0.1-1.0-Mild gingivitis 1.1-2-Moderate gingivitis 2.1-3.0 Severe gingivitis
VAS score | Changes from baseline to 7th day, 14th day, 21st day and 28th day
  Index given by Freyd in 1923 Scale -1-10 Score Scale: 0-10 Score 0-No pain 1-3: Mild 4-6: Moderate 7-9: severe 10-worst

IPD SHARING:
Plan to Share IPD: No
For the purpose of confidentiality as will be promised to the participants while signing the informed consent , all individual records except that of the parameters assessed during the study and the photographs taken will remain unshared to the public or fellow researchers